CLINICAL TRIAL: NCT05312515
Title: The Effect of Hot Bag/Warm Application on Feet After Cesarean Delivery on Postpartum Comfort, Pain and Flatus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Yasemin ERKAL AKSOY, Asistant Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0000-0002-7453-1205
Record Dates: First submitted 2022-03-23; First posted 2022-04-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cesarean Section Complications; Pain; Postpartum Anxiety
Keywords: Cesarean Section; Pain; Postpartum Comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In order to ensure randomization in the study, a random numbers table was created by dividing into two groups out of 238 samples by taking 10% more than the number of samples determined on the site https://www.randomizer.org/. In order to avoid bias, the assignment of women to the intervention and control groups according to the randomization list will be determined by a midwife working in the clinic, who is not one of the study authors. In the study, the CONSORT scheme will be followed during the application.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Application to Feet and Follow-up After Cesarean Section (Experimental): Warm application will be applied to the feet of women who come to the surgical service after cesarean delivery, 3 hours after they are admitted to the service. For hot application, a hot water bag will be used, the temperature of the water to be placed in the hot water bag is max. It will be set by the researcher to be 44°C. Since the temperature of the water (max. 44°C) does not create a risk of burns, no additional precautions were required. A stopwatch clock will be used to track the duration of the application. After the application will be done for 30 minutes, a hot water bag will be taken. Hot application will be done once. During the application, the researcher will be with the women, will check whether any complications have developed, and if complications or discomfort develop, the application will be terminated.
  Interventions: Other: Warm Application to Feet
- Control (No Intervention): The control group will be given routine post-operative care without any intervention and data collection tools will be applied at the same time as the intervention group. In addition, the patient and his family will be informed to write it down with the watch if there is gas after the procedure when the researcher is not with them.

INTERVENTIONS:
Other: Warm Application to Feet — Warm Application to Feet after Cesarean Section
  Arms: Warm Application to Feet and Follow-up After Cesarean Section

SUMMARY:
The postpartum period is a process in which both physical (bleeding, infection, anemia) and emotional (delay in breastfeeding and mother-baby relationship) problems occur in women. Among the conditions that physically affect the woman who has had a cesarean section, a decrease in bowel movements is often seen and this decrease can last for 24 hours or longer. Initiation of bowel movements after surgery, time of first flatulence and defecation are important factors that determine postoperative patient comfort.

DETAILED DESCRIPTION:
Pain after cesarean section is usually associated with incision site and uterine contractions. There are various medical treatment and midwifery applications for the resolution of pain and gas output after cesarean section. Recently, it has been stated that in addition to the treatments applied after surgery, non-drug methods should be used to increase the effectiveness of recovery. These methods include applications such as hot application, abdominal massage, music therapy, chewing gum. The effect of hot application in patients with post-operative gas problems is the acupuncture points of the foot, warm and moist heat stimulation and the small intestine, colon, anus and other reflective areas. activates blood circulation. It is predicted that postpartum comfort will increase in the postpartum postpartum, whose pain decreases with postpartum heat application and intestinal mobility returns to normal. The aim of this study is to determine the effect of applying heat to the feet after cesarean section on postpartum comfort, pain and gas output.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Can read and understand Turkish
* No history of any medical illness
* Singular pregnancy
* No complications during or after surgery
* Those who have not had any problems during pregnancy
* giving birth to a live baby
* No diagnosed psychological disorder
* Women who do not pass gas before applying heat

Exclusion Criteria:

* From gas before hot application
* Hearing loss
* The baby is in intensive care
* Women with vascular diseases
* Women who were taken to the intensive care unit after surgery due to any complications

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 108 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | at the beginning of the study
  It was prepared by the researcher to describe the sociodemographic characteristics and current health status of women. The group of women will be marked as Intervention or Control.
Post Cesarean Section Follow-up Form-First follow up | application after 30 minute
  In this form, the time the patient was taken into surgery; length of stay in the recovery unit; time of service; the type of anesthesia administered; It was created by the researcher in order to obtain information about the hot water bag application time and the first gas removal time.
Post Cesarean Section Follow-up Form-Second follow up | application after 60 minute
  In this form, the time the patient was taken into surgery; length of stay in the recovery unit; time of service; the type of anesthesia administered; It was created by the researcher in order to obtain information about the hot water bag application time and the first gas removal time.
Post Cesarean Section Follow-up Form-Third follow up | application after 120 minute
  In this form, the time the patient was taken into surgery; length of stay in the recovery unit; time of service; the type of anesthesia administered; It was created by the researcher in order to obtain information about the hot water bag application time and the first gas removal time.

SECONDARY OUTCOMES:
Visual Pain Scale (VAS)-First follow up | application after 30 minute
  It is a measurement usually used to evaluate pain from 0 (no pain) to 10 (unbearable pain). In this assessment scale, the patient is asked to express the level of pain he/she feels at that moment with numbers. The number expressed by the patient is accepted as the intensity of pain felt at that moment.
Visual Pain Scale (VAS)-Second follow up | application after 60 minute
  It is a measurement usually used to evaluate pain from 0 (no pain) to 10 (unbearable pain). In this assessment scale, the patient is asked to express the level of pain he/she feels at that moment with numbers. The number expressed by the patient is accepted as the intensity of pain felt at that moment.
Visual Pain Scale (VAS)-Third follow up | application after 120 minute
  It is a measurement usually used to evaluate pain from 0 (no pain) to 10 (unbearable pain). In this assessment scale, the patient is asked to express the level of pain he/she feels at that moment with numbers. The number expressed by the patient is accepted as the intensity of pain felt at that moment.
Postpartum Comfort Scale-First follow up | application after 30 minute
  Postpartum Comfort Scale: It is a scale that can be used to measure the postpartum comfort of mothers who delivered vaginally or by cesarean section. The PCS consists of a 5-point Likert-type scale scoring system and 34 items. I totally agree with positive sentences shows the best comfort (5 points), and negative sentences show low comfort (1 point). Accordingly, the lowest score to be taken from the scale is 34, and the highest score is 170. The average value is determined by dividing the total score obtained from the scale by the number of items, and the result is shown in the 1-5 distribution.High scores on the scale indicate increased comfort.
Postpartum Comfort Scale -Second follow up | application after 60 minute
  Postpartum Comfort Scale: It is a scale that can be used to measure the postpartum comfort of mothers who delivered vaginally or by cesarean section. The PCS consists of a 5-point Likert-type scale scoring system and 34 items.I totally agree with positive sentences shows the best comfort (5 points), and negative sentences show low comfort (1 point). Accordingly, the lowest score to be taken from the scale is 34, and the highest score is 170. The average value is determined by dividing the total score obtained from the scale by the number of items, and the result is shown in the 1-5 distribution.High scores on the scale indicate increased comfort.
Postpartum Comfort Scale -Third follow up | application after 120 minute
  Postpartum Comfort Scale: It is a scale that can be used to measure the postpartum comfort of mothers who delivered vaginally or by cesarean section. The PCS consists of a 5-point Likert-type scale scoring system and 34 items. I totally agree with positive sentences shows the best comfort (5 points), and negative sentences show low comfort (1 point). Accordingly, the lowest score to be taken from the scale is 34, and the highest score is 170. The average value is determined by dividing the total score obtained from the scale by the number of items, and the result is shown in the 1-5 distribution. High scores on the scale indicate increased comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ali Kemal Belviranlı Gynecology and Pediatrics Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Büyükkayacı Duman N, Karataş N. Sezaryen Sonrası Erken Taburcu Olan Kadınlara Verilen Evde Bakım Hizmetinin Anne Sağlığına Ve Öz Bakım Gücüne Etkisi. Sağlık Bil Derg 2011, 20(1):54-67.
- [Background] Ciardulli A, Saccone G, Di Mascio D, Caissutti C, Berghella V. Chewing gum improves postoperative recovery of gastrointestinal function after cesarean delivery: a systematic review and meta-analysis of randomized trials. J Matern Fetal Neonatal Med. 2018 Jul;31(14):1924-1932. doi: 10.1080/14767058.2017.1330883. Epub 2017 Jun 6. PMID 28502203
- [Background] Sutton CD, Carvalho B. Optimal Pain Management After Cesarean Delivery. Anesthesiol Clin. 2017 Mar;35(1):107-124. doi: 10.1016/j.anclin.2016.09.010. Epub 2016 Dec 12. PMID 28131114
- [Result] Sell SE, Beresford PC, Dias HHZR, Garcia ORZ, Santos EKA. Looks and knowledge: experiences of mothers and nursing staff regarding post-caesarean section pain. Text Context Nurs., 2012, 21(4): 766-74.